CLINICAL TRIAL: NCT07154225
Title: INcreasing Adolescent Social and Community SupporT - Full Trial
Acronym: INACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Manchester (Other); National Academy for Social Prescribing (Unknown); We Do Wellbeing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1207
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Loneliness
Keywords: Loneliness; Social Prescribing; Schools; Pupils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Prescribing (Experimental): SP is a person-centred approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and Link Workers (LWs), based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have a good knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioural activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that best match their preferences.
  Interventions: Behavioral: Social Prescribing
- Signposting (Active Comparator): Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of school pastoral staff meeting with YP identified as lonely and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Interventions: Behavioral: Signposting

INTERVENTIONS:
Behavioral: Social Prescribing — SP is a person-centred approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and Link Workers (LWs), based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have a good knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioural activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that best match their preferences.
  Arms: Social Prescribing
Behavioral: Signposting — Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of school pastoral staff meeting with YP identified as lonely and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Arms: Signposting

SUMMARY:
Background: Social Prescribing is a mechanism of connecting patients with non-medical forms of support within the community and has been shown to improve loneliness. Yet update from young people has been lower than for adults. This is thought to be due to accessibility issues as young people are less likely to draw on primary care, where social prescribing is based, for wellbeing support. The INACT pilot sought to test the feasibility and acceptability of a Social Prescribing pathway via schools to support young people who are lonely through a randomised controlled trial. Findings suggested that study procedures, including the measures were appropriate and that Social Prescribing was deemed by young people, social prescribers and school staff as feasible, acceptable and suitable and there was evidence of impact in the social prescribing arm when compared to signposting. Given the positive pilot findings, the aim of the INACT full trial is to build upon the pilot work and conduct a clinical and cost effectiveness trial into the impact of Social Prescribing in schools for loneliness and low community connection, compared to signposting.

Methods: A minimum of 215 pupils reporting loneliness will be recruited across 30 mainstream schools in England and be randomly allocated to signposting or Social Prescribing. Pupils in the control group will receive signposting to sources of support from school staff. The co-produced social prescribing intervention includes up to 6 sessions with a Link Worker who will work with individuals to understand 'what matters to them' and connect them with local sources of support. The clinical and cost effectiveness of Social Prescribing for young people with loneliness will be assessed using measures of loneliness, mental health, wellbeing, quality of life, and service use. Data will be collected at baseline and 3, 6, and 12 months later. Qualitative interviews will also be conducted to explore barriers, facilitators, mechanisms of change and impact.

Discussion: INACT will provide evidence of the clinical and cost effectiveness of Social Prescribing in schools for supporting young people experiencing loneliness. It will also establish what types of community and social activities young people engage in and what factors affect participation.

ELIGIBILITY:
Inclusion Criteria

1. Schools:

   * A primary or secondary school willing to participate in INACT
   * In England
   * Have classes of pupils in eligible year groups to participate (Years 5, 7, 8)
2. Pupils and their parents/guardians:

   * Score 7 or above on the Good Childhood Index (indicating high loneliness)
   * Parents/guardians consent, and pupils assent, to get support

Exclusion Criteria

1. Schools:

   * Private schools or sixth form/colleges
   * Specialist schools
   * Schools only offering alterative provision
   * Outside of England
   * Does not have classes of pupils in eligible year groups to participate (Years 4, 5, 7, 8)
2. Pupils and their parents/guardians:

   * Score below 7 on the Good Childhood Index (indicating low loneliness)
   * Parents/guardians do not consent, or pupils do not assent, to get support
   * Children and young people with severe learning disabilities who are unable to complete questionnaires

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Baseline, 3, 6 and 12 months
  Measured using the Good Childhood Index containing 3 questions on a 3-point Likert scale (scoring between 3-9). Higher scores indicate higher reported loneliness. Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
Wellbeing | Baseline, 3, 6 and 12 months
  Measures using the Wellbeing subscale (Kidscreenn-52) which contains 6 questions each on a five-point Likert scale (scoring between 6-30). Higher scores indicate greater well-being.
Mental health (emotional difficulties) | Baseline, 3, 6 and 12 months
  Measured using the Emotional difficulties subscale (Me and My feelings questionnaire) which contains 10 questions on a 3-point Likert scale (scoring between 0-20). Higher scores indicate higher emotional difficulties.
Service use | Baseline, 3, 6 and 12 months
  Measures using the Client Service Receipt of Inventory which contains 11 questions on a five-point Likert scale. Scoring can be looked at by individual items (i.e. score between 1-5) or by scoring all items (i.e. scores between 11-55). Higher scores indicate more contact with a service/services.
Quality of Life | Baseline, 3, 6 and 12 months
  Measured using the CHU-9D which contains 9 questions on a five-point Likert scale (scoring between 1-5). Higher scores indicate higher quality of life.
Stress | Baseline, 3, 6 and 12 months
  Measured using the Perceived Stress Scale 4 which assesses stress using 4 questions on a five-point Likert scale (scoring between 0-16). Higher scores indicate higher levels of perceived stress (secondary school pupils only)
Emotion Regulation | Baseline, 3, 6 and 12 months
  Emotion Regulation Index for Children and Adolescents is assessed using 16 items on a five-point Likert scale (scoring between 1-5). Higher scores indicate greater emotion regulation.
Intervention Acceptability | 3, 6, and 12 months
  Measured using a single item adapted from the NHS Friends and Family Test on a five-point Likert scale . Higher scores indicate higher acceptability. Social prescribing arm only.
Intervention Feasibility (School Staff and Link Workers), | Approx 3 months after intervention delivery has begun
  Measured using the Feasibility of Intervention Measure (FIM) which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention feasibility.
Intervention Acceptability (School Staff and Link Workers) | Approx 3 months after intervention delivery has begun
  Measured using the Acceptability of Intervention Measure (AIM) which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention acceptability.
Intervention Appropriateness (School Staff and Link Workers) | Approx 3 months after intervention delivery has begun
  Measured using the Intervention Appropriateness Measure (IAM) which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention appropriateness. 3 months

OTHER OUTCOMES:
Family Support | Baseline, 3, 6 and 12 months
  Measured using The Family Support Subscale (Student Resilience Survey) which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher family support.
School Support | Baseline, 3, 6 and 12 months
  Measured using The School Support Subscale (Student Resilience Survey) which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher school support.
Problem Solving | Baseline, 3, 6 and 12 months
  Measured using The Problem Solving subscale (Student Resilience Survey) which contains 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher problem solving with others.
Social support subscale | Baseline, 3, 6 and 12 months
  Measured using the CYRM-R which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher social support.
Local environment | Baseline, 3, 6 and 12 months
  Measured using the HBSC 2022 which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate a more positive view of ones local environment.
Activity Engagement | Baseline, 3, 6 and 12 months
  Measured using the BeeWell survey which contains 11 questions each on a six-point Likert scale (scoring between 11-66). Higher scores indicate higher daily engagement with more activities. Each item can also be scored individually and indicates more frequent engagement with that activity.
Bullying (primary school pupils) | Baseline, 3, 6 and 12 months
  Measured using the Bullying subscale (Kidscreen 52) which contains 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher levels of bullying.
Bullying (secondary school pupils) | Baseline, 3, 6 and 12 months
  Measured using the BeeWell survey which contains 3 questions each on a four-point Likert scale (scoring between 0-9). Higher scores indicate higher levels of bullying.
Social structure and quality | Baseline, 3, 6 and 12 months
  Measured using 5 questions adapted from PISA 2022 and MCS4. One of which requires an open-ended numerical value and four questions which are rated on a five-point Likert scale (scoring between 0-16). Higher scores indicate a greater social structure and friendship quality.
Flow | Baseline, 3, 6 and 12 months
  Measured using using The General Flow Proneness Scale (secondary school pupils only) which consists of 13 questions each on a five-point Likert scale (scoring between 13-65). Higher scores indicate higher flow experience.
Therapeutic Alliance (Social Prescribing arm) | 3, 6 and 12 months
  Measured using the Session Feedback Questionnaire which contains 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher therapeutic alliance.

IPD SHARING:
Plan to Share IPD: Undecided
Some IPD data will be shared but specific data is being currently discussed with the funder. We will update this record when we know more.